CLINICAL TRIAL: NCT00224471
Title: A Phase III, Double-blind, Randomized, Study to Compare: 1) the Immunogenicity and Safety of 3 Commercial Scale Consistency Lots of GlaxoSmithKline (GSK) Biologicals' Herpes Simplex Candidate Vaccine in Healthy HSV-1 and -2 Seronegative (HSV 1-/2-) Female Subjects Aged 10 - 17 Years, and 2) Vaccine Immunogenicity in Healthy HSV 1-/2- Females Aged 10 - 17 Years With Healthy HSV 1-/2- Adult Females
Brief Title: Study to Compare Safety and Immunogenicity of Commercial Scale Consistency Lots of Herpes Simplex Vaccine
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 208141/042
Record Dates: First submitted 2005-09-21; First posted 2005-09-23 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Herpes Simplex
Keywords: Adolescents; Immunogenicity; Safety; Herpes Simplex vaccine
MeSH Terms: conditions — Herpes Simplex | interventions — Herpes Simplex Virus Vaccines

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Group A (Experimental)
  Interventions: Biological: GSK208141 vaccine
- Group B (Experimental)
  Interventions: Biological: GSK208141 vaccine
- Group C (Experimental)
  Interventions: Biological: GSK208141 vaccine

INTERVENTIONS:
Biological: GSK208141 vaccine — 3 IM doses
  Other Names: Herpes simplex vaccine

SUMMARY:
Evaluate, one month after the third dose, the lot-to-lot consistency of 3 different commercial scale production lots of the candidate vaccine in healthy HSV 1-/2- females aged 10-17 years, determined by ELISA. Absence in significant variation for both parameters among the tested lots was hypothesized.

DETAILED DESCRIPTION:
At month 0, 1 and 6, 3 groups of 184 subjects received each 3 doses of herpes simplex vaccine lot A, B or C, respectively. The study took 14 months to complete, including screening, and 6 visits were required. The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Healthy female between, and including, 10 and 17 years of age at the time of the first vaccination.
* Seronegative for HSV-1 and HSV-2 at screening
* Written informed assent obtained from the subject and written informed consent obtained from a parent or legal guardian of the subject prior to enrolment. If the subject is above the legal age of consent in her country, written informed consent will only be obtained from the subject.
* Subject must have a negative urine pregnancy test.
* Subject must be of non-childbearing potential, i.e. pre-menarcheal, or if of childbearing potential she must be abstinent or must be using an effective method of birth control for 30 days prior to vaccination, have a negative urine pregnancy test and must agree to continue such precautions for two months after completion of the vaccination series. Subjects who reach menarche during the study and therefore are of childbearing potential must agree to follow the same precautions.
* A subject who (or whose parents/guardian) the investigator believes can and will comply with the requirements of the protocol

Exclusion criteria:

* Pregnant or lactating female.
* Female planning to become pregnant during the first eight months of the study
* Any previous history of, or current clinical signs or symptoms of oro-labial (cold sores), genital or non-genital HSV disease, such as swelling, papules, vesicles, pustules, ulcers, crusts, fissures, erythema, discharge, pain, burning, itching, tingling, or dysuria.
* Previous vaccination against herpes.
* History of erythema multiforme.
* Use of any investigational or non-registered drug or vaccine other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Planned administration/administration of a non-study vaccine within 30 days before and after the first dose of study vaccine with the following exceptions: Administration of routine meningococcal, hepatitis B, inactivated influenza, diphtheria/tetanus and/or diphtheria/tetanus containing vaccine up to 8 days before the first dose of study vaccine is allowed.
* History of allergic disease or reactions likely to be exacerbated by any component of the study vaccines
* Any confirmed or suspected immunosuppressive or immunodeficient condition, including human immunodeficiency virus (HIV) infection.
* History of a current acute or chronic autoimmune disease.
* History of any neurologic disorders or seizures, with the exception of a single febrile seizure during childhood.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by medical history or physical examination.
* Acute disease at the time of enrolment
* Oral temperature ≥99.5°F (> 37.5°C) / axillary temperature ≥99.5°F (> 37.5°C) at the time of enrolment
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs within six months prior to the first vaccine dose or planned use during the study period
* Administration of immunoglobulins and/or any blood products within the three months preceding the first dose of study vaccine or planned administration during the study period.

Ages: 10 Years to 17 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 671 (Actual)
Dates: Start 2003-12; Primary Completion 2005-09 (Actual); Study Completion 2006-01 (Actual)

PRIMARY OUTCOMES:
Anti-gD antibody titre in the entire cohort (10-17 yrs) | At month 7

SECONDARY OUTCOMES:
Anti-gD antibody titre | At months 2 and 12
Anti-HSV neutralizing antibodies | At months 2, 7 and 12
Occurrence and intensity of solicited local symptoms. Resulting school absenteeism will also be evaluated. | Within 7 days after each vaccination
Occurrence, intensity, relationship to vaccination and resulting school absenteeism of solicited general symptoms | Within 7 days after each vaccination
Occurrence, intensity, relationship to vaccination and resulting school absenteeism of unsolicited adverse events | Within 30 days after any vaccination
Occurrence of new onset chronic diseases and other medically significant conditions, regardless of causal relationship to vaccination and intensity | Throughout the study
Occurrence and relationship to vaccination of SAEs | Throughout the study period
Anti-gD antibody titre in sera from HSV-042 subjects and in an equally sized subset of sera from adults from study 208141/039 | At month 7
Seroconversion rate by anti-gD ELISA. in HSV-042 subjects and in an equally sized subset of adults from study 208141/039 | At month 7
In the event that a cell-mediated immune correlate of protection is identified in study 208141/039: assessment of the immune correlate of protection in a random subset of HBV-042 subjects | At months 0, 2, 7, and 12

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (12):
- United States (8):
  - GSK Investigational Site, Mesa, Arizona
  - GSK Investigational Site, Fountain Valley, California
  - GSK Investigational Site, Golden, Colorado
  - GSK Investigational Site, Cincinnati, Ohio
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Galveston, Texas
  - GSK Investigational Site, Salt Lake City, Utah
  - GSK Investigational Site, Seattle, Washington
- GSK Investigational Site, Ghent, Belgium
- Canada (3):
  - GSK Investigational Site, Edmonton, Alberta
  - GSK Investigational Site, Vancouver, British Columbia
  - GSK Investigational Site, Beauport, Quebec

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: 208141/042 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 208141/042 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 208141/042 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 208141/042 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 208141/042 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 208141/042 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register